CLINICAL TRIAL: NCT03842501
Title: A Randomized, Double-blind, Placebo-controlled Study Evaluating the Effects of the GOLO Weight Management Program With and Without Release Supplement on Weight and Metabolic Parameters in Subjects With Obesity
Brief Title: Effects of the GOLO Weight Management Program With and Without Release Supplement on Weight and Metabolic Parameters in Subjects With Obesity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Golo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GOLO1703
Record Dates: First submitted 2019-02-13; First posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- Release supplement (Experimental)
  Interventions: Dietary Supplement: Release Supplement

INTERVENTIONS:
Dietary Supplement: Release Supplement — Calorie reduced diet plus Release supplement
  Arms: Release supplement
Dietary Supplement: Placebo — Calorie reduced diet plus Placebo
  Arms: Placebo

SUMMARY:
This randomized, double-blind placebo-controlled study was intended to measure the effects of the GWMP with Release supplement versus GWMP with placebo supplement in a representative group of obese subjects with or without diabetes at one outpatient medical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years and ≤ 80 years
2. Body mass index (BMI) ≥ 30 and ≤ 60 kg/m2
3. Have the ability to engage in at least 15 minutes of moderate physical activity such as brisk walking
4. Willing to comply with study procedures described herein

Exclusion Criteria:

1. Current diagnosis of type 1 diabetes
2. Subjects with a history of hypoglycemia
3. A history of an eating disorder as defined by the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5)
4. Known allergy to any of the components in the Release supplement
5. A history of prior surgery for weight loss
6. Currently taking injectable medications to control diabetes, including insulin and GLP-1 agonists
7. Currently pregnant or breastfeeding or have had a baby within the last six weeks
8. Planning to become pregnant in the next three months. Women of child bearing potential must be willing and able to use adequate and reliable contraception throughout the study (e.g. abstinence or barrier with additional spermicidal foam or jelly, or the use of intrauterine device or hormonal contraception).
9. Uncontrolled hypertension at screening defined as Systolic blood pressure greater than 180 mmHG or Diastolic blood pressure greater than 110 mmHG
10. Current clinical diagnosis or signs and symptoms of unstable (in the opinion of the principle investigator) heart, kidney or liver disease, cancer, or chronic neurological disease.
11. Current participation in any other weight loss or weight management program
12. Currently taking weight loss medications, or medications or supplements known to be associated with significant weight loss or weight gain
13. Has any condition that, in the opinion of the investigator, would make participation in this study not in the best interest of the subject or that could prevent, limit or confound the protocol-specified assessments. Examples include: history of diabetic ketoacidosis; active chronic liver disease or cirrhosis; chronic autoimmune disease; inflammatory bowel disease, colonic ulceration, partial intestinal obstruction, subjects predisposed to intestinal obstruction; chronic intestinal diseases associated with marked disorders of digestion or absorption

    -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2018-12-24 (Actual); Study Completion 2018-12-24 (Actual)

PRIMARY OUTCOMES:
Change in weight from baseline | 13 weeks

SECONDARY OUTCOMES:
Change in waist circumference from baseline | 13 weeks
Change in fasting glucose from baseline | 13 weeks
Change in Hemoglobin A1C from baseline | 13 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Buynak Clinical Research, Valparaiso, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided